CLINICAL TRIAL: NCT03323606
Title: Online Interventions for Problem Gamblers With and Without Co-occurring Problem Drinking: Randomized Controlled Trial
Brief Title: Online Interventions for Gamblers With and Without Co-occurring Problem Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University of Calgary (Other); University of Manitoba (Other)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 010/2017
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Gambling; Alcohol Consumption
MeSH Terms: conditions — Gambling; Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gambling Internet Intervention (Active Comparator): The gambling only Internet intervention (G-only) will consist of a new online version of self-change tools that have previously been translated successfully into an online form and shown to have a significant impact on gambling in three trials. A major focus of this intervention is to provide individuals with clear and concise behavioral and cognitive strategies for meeting the goal of reducing or quitting gambling.
  Interventions: Behavioral: Gambling Internet Intervention
- Gambling Internet Intervention + CYD (Experimental): The G+A intervention condition will consist of the G-only intervention and an online intervention for drinking. The online drinking intervention chosen is Check Your Drinking, a brief online intervention designed to provide personalized normative feedback aimed at motivating reductions in drinking
  Interventions: Behavioral: Gambling Internet Intervention; Behavioral: Check Your Drinking

INTERVENTIONS:
Behavioral: Gambling Internet Intervention — The gambling Internet intervention consists of a new online version of self-change tools that have previously been translated successfully into an online form and shown to have a significant impact on gambling in three trials. A major focus of this intervention is to provide individuals with clear and concise behavioral and cognitive strategies for meeting the goal of reducing or quitting gambling.
Behavioral: Check Your Drinking — A brief online intervention designed to provide personalized normative feedback aimed at motivating reductions in drinking
  Arms: Gambling Internet Intervention + CYD

SUMMARY:
Many problem gamblers are also problem drinkers,with lifetime prevalence in nationally representative samples ranging from 45% to 73%. Heavy drinking often occurs while problem gamblers are engaging in gambling activities, resulting in increased risky gambling behaviour. Further, co-occurring problem drinking negatively impacts on the treatment outcomes of problem gamblers. Thus, targeting problem drinking among problem gamblers may have the dual benefits of reducing both the problem drinking itself, and of acting as a mediator for reductions in problem gambling behaviour. The present study seeks to determine whether providing simultaneous access to help for gambling and drinking is of benefit for those with these co-occurring problems.

DETAILED DESCRIPTION:
Problem gambling and problem drinking frequently co-occur. Further, the treatment needs of people with co-occurring gambling and drinking problems may be different from those of problem gamblers who do not drink alcohol in a hazardous fashion. The current project will evaluate whether there is a benefit to providing access to a problem drinking Internet intervention (G+A intervention) in addition to an Internet intervention for problem gambling (G-only intervention) in participants with gambling problems who do or do not have co-occurring problem drinking.

People with gambling concerns will be recruited using targeted advertisements. Potential participants will be screened using an online survey to identify participants meeting criteria for problem gambling. As part of the baseline screening process, measures of alcohol consumption will be assessed. Eligible participants who agree to take part in the study will be randomized into one of two online interventions for gamblers - an intervention that only targets gambling issues (G-only) versus one that contains an intervention for drinking (G+A). It is predicted that for problem gamblers with co-occurring problem drinking, participants provided access to the G+A website will display significantly reduced gambling outcomes at three- and six-month follow-ups as compared to those provided access to the G-only website. However, for problem gamblers without co-occurring problem drinking, it is predicted that participants will display no significant difference between the G-only and G+A websites at three- and six-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* Score of 3 or greater on the Problem Gambling Severity Index of the Canadian Problem Gambling Index (PGSI- CPGI)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
The NORC DSM-IV Screen for Gambling Problems (NODS) past 3 month version indicating DSM-IV gambling severity. | 3 and 6 months
  Change in gambling severity (NODS) from baseline
Number of days gambled per month | 3 and 6 months
  Change in mean days per month gambling from baseline

CONTACTS AND LOCATIONS:
Overall Officials: John A Cunningham, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cunningham JA, Hodgins DC, Keough M, Hendershot CS, Schell C, Godinho A. Online interventions for problem gamblers with and without co-occurring unhealthy alcohol use: Randomized controlled trial. Internet Interv. 2020 Jan 18;19:100307. doi: 10.1016/j.invent.2020.100307. eCollection 2020 Mar. PMID 32042600
- [Derived] Cunningham JA, Hodgins DC, Keough M, Hendershot CS, Bennett K, Bennett A, Godinho A. Online interventions for problem gamblers with and without co-occurring problem drinking: study protocol of a randomized controlled trial. Trials. 2018 May 25;19(1):295. doi: 10.1186/s13063-018-2672-x. PMID 29801520
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research